CLINICAL TRIAL: NCT02711904
Title: Effect of Two Plasma Concentrations of Remifentanil Through Target Controlled Anesthesia on Frequency and Intensity of Coughing During Extubation: Randomized Controlled Clinical Trial
Brief Title: Concentrations of Remifentanil for Extubation
Acronym: REMEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seganest (Other)
Collaborators: Instituto Para Ninos Ciegos y Sordos del Valle del Cauca (Other)
Responsible Party: Principal Investigator, LUIS ALBERTO TAFUR B, Principal Investigator, Seganest
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SEGANEST
Record Dates: First submitted 2013-08-27; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Cough
Keywords: Extubation; Cough; Target Controlled Anesthesia (TACAN)
MeSH Terms: conditions — Cough | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extubation U (Active Comparator): Remifentanil concentration between 2 - 3 ng/ml.
  Interventions: Drug: Extubation U
- Extubation T (Experimental): Remifentanil concentration between 3 - 4 ng/ml
  Interventions: Drug: Extubation T

INTERVENTIONS:
Drug: Extubation U — Dose of remifentanil according to the randomization; the infusions that were used to reach the PC target were:
  * 20 years old - 6.0 mcg/Kg/h
  * 30 years old - 5.7 mcg/Kg/h
  * 40 years old - 5.3 mcg/kg/h
  * 50 years old - 5.0 mcg/kg/h
  * 60 years old - 4.6 mcg/kg/h
  * 70 years old - 4.3 mcg/kg/h
  * 80 years old - 4.0 mcg kg/h.
  Other Names: Ultiva
  Arms: Extubation U
Drug: Extubation T — Dose of infusion of remifentanil to reach a PC 3 - 4 ng/ml, in the following manner:
  The assistant placed the infusion balloon in such a way that it could not be seen by the treating anesthesiologist, he proceeded to open the corresponding wrapping according to the consecutive which corresponds to the patient.
  The remifentanil dose was adjusted according to the randomization:
  * 20 years old - 9.0 mcg/Kg/h
  * 30 years old - 8.5 mcg/Kg/h
  * 40 years old - 8.0 mcg/kg/h
  * 50 years old - 7.5 mcg/kg/h
  * 60 years old - 7.0 mcg/kg/h
  * 70 years old - 6.5 mcg/kg/h
  * 80 years old - 6.0 mcg kg/h.
  Other Names: Ultiva
  Arms: Extubation T

SUMMARY:
Condition of the State: (terminated, recruiting, etc.) Terminated

Study Design: Main Objective:

Compare the frequency and intensity of coughing at the time of extubation with two infusions of remifentanil that predict a plasma concentration (PC) of 3 - 4 and 2 - 3 ng/ml, through the technique of target controlled anesthesia

DETAILED DESCRIPTION:
Phase of the study:

Phase IV

Intervention:

Drug: U Extubation

Other Names:

Concentration 2 - 3 ng/ml Dose of remifentanil according to the randomization: Letter U between 2 - 3 ng/ml. The infusions that were used to reach the (PC) target were: Group U = 2 - 3 ng/ml. 20 years old - 6.0 mcg/Kg/h, 30 years old - 5.7 mcg/Kg/h, 40 years old - 5.3 mcg/kg/h, 50 years old - 5.0 mcg/kg/h, 60 years old - 4.6 mcg/kg/h, 70 years old - 4.3 mcg/kg/h, 80 years old - 4.0 mcg kg/h.

Drug: Extubation T

Other Names:

Concentration 3 - 4 ng/ml Dose of infusion of remifentanil to reach a (PC) 3 - 4 ng/ml, in the following manner: The assistant placed the infusion balloon in such a way that it could not be seen by the treating anesthesiologist, he proceeded to open the corresponding wrapping according to the consecutive which corresponds to the patient. The remifentanil dose was adjusted according to the randomization: Group T = 3 - 4 ng/ml. 20 years old - 9.0 mcg/Kg/h, 30 years old - 8.5 mcg/Kg/h, 40 years old - 8.0 mcg/kg/h, 50 years old - 7.5 mcg/kg/h, 60 years old - 7.0 mcg/kg/h, 70 years old - 6.5 mcg/kg/h, 80 years old - 6.0 mcg kg/h.

Number of arms:

2

Masking:

The patient had masking with regards to the anesthetic procedure from the unfamiliarity per se of the same and by agents used in this that induced anxiolysis and hypnosis.

To guarantee the masking to the viewer, which was the treating anesthesiologist, a nurse was trained in the adjustment of the infusion balloon. Ten minutes before concluding the procedure and by request of the anesthesiologist, the nurse proceeded to locate balloon in such a way that the infusion could not be seen by the anesthesiologist, then opened the envelope and adjusted the infusion according to the randomization (U) o (T). The evaluation of the cough, its intensity and the Ramsay were under the care of the anesthesiologist, who was unaware of the awakening infusion.

Allocation:

Two were allocated for the use: Concentration of remifentanil of 2 - 3 ng/ml (group U) and concentration of remifentanil of 3 - 4 ng/ml (group T).

Recruitment:

A patient was recruited between the period of January 2011 and July 2012.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18-70 years
* Risk Scale American Society of Anaesthesiologists physical status classification (ASA) I and II
* Undergoing elective ear surgery

Exclusion Criteria:

* Patients who are contraindicated remifentanil
* Patients undergoing emergency surgery
* Pulmonary Pathology (ASTHMA - COPD)
* Index of body mass greater than 35
* Background of respiratory failure three weeks prior to the procedure
* Smokers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Cough | It is evaluated by the scale of cough over a two hour period after surgery: is assessed at 5 minutes turned off the halogenated inhalation anesthetics, thereafter every minute until the patient responds to verbal stimulus and can be extubated
  Number of episodes and duration of cough that occur when the patient responds to verbal stimulus and extubated.
  Cough Scale
  * Grade 0 = No cough
  * Grade 1 = Mild (only episode of cough)
  * Grade 2 = Moderate (more than 1episode of cough during less than 5 seconds)
  * Grade 3 = Severe (More than one episode of cough that lasted more than 5 seconds or purposeless movements of the extremities).

SECONDARY OUTCOMES:
Wake time. | During two hours after surgery, five minutes after turning off halogenated inhaled anesthetics, then every minute until the patient opens his eyes and is extubated.
  When vaporizer where closed until the patient responds to the verbal stimulus and is extubated.
  Defined as the time taken to open eyes after having turned off the halogenated inhalation anesthetics.
Ramsay scale at the time of extubation | During two hours after surgery, the estimated time period during which the event was assessed five (5) minutes after every minute, until answered
  Ramsay scale: score objective system for measuring drug-induced sedation
  * Score 1: Anxious or restless or both
  * Score 2: Cooperative, orientated and tranquil
  * Score 3: Responding to commands
  * Score 4: Brisk response to stimulus
  * Score 5: Sluggish response to stimulus
  * Score 6: No response to stimulus

CONTACTS AND LOCATIONS:
Overall Officials: LUIS A TAFUR, MD, Principal Investigator — Seganest; Eduardo Lema, MD, Study Director — Seganest
Locations (1):
- Instituto Para Niños Ciegos y Sordos del Valle del Cauca, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No
The individual data of the participants (IPD) were only available to the ethics committee of the institution.

REFERENCES:
- [Background] Neelakanta G, Miller J. Minimum alveolar concentration of isoflurane for tracheal extubation in deeply anesthetized children. Anesthesiology. 1994 Apr;80(4):811-3. doi: 10.1097/00000542-199404000-00013. PMID 8024135
- [Background] Guler G, Akin A, Tosun Z, Eskitascoglu E, Mizrak A, Boyaci A. Single-dose dexmedetomidine attenuates airway and circulatory reflexes during extubation. Acta Anaesthesiol Scand. 2005 Sep;49(8):1088-91. doi: 10.1111/j.1399-6576.2005.00780.x. PMID 16095449
- [Background] Saghaei M, Reisinejad A, Soltani H. Prophylactic versus therapeutic administration of intravenous lidocaine for suppression of post-extubation cough following cataract surgery: a randomized double blind placebo controlled clinical trial. Acta Anaesthesiol Taiwan. 2005 Dec;43(4):205-9. PMID 16450594
- [Background] Minogue SC, Ralph J, Lampa MJ. Laryngotracheal topicalization with lidocaine before intubation decreases the incidence of coughing on emergence from general anesthesia. Anesth Analg. 2004 Oct;99(4):1253-1257. doi: 10.1213/01.ANE.0000132779.27085.52. PMID 15385385
- [Background] Fagan C, Frizelle HP, Laffey J, Hannon V, Carey M. The effects of intracuff lidocaine on endotracheal-tube-induced emergence phenomena after general anesthesia. Anesth Analg. 2000 Jul;91(1):201-5. doi: 10.1097/00000539-200007000-00038. PMID 10866913
- [Background] Tagaito Y, Isono S, Nishino T. Upper airway reflexes during a combination of propofol and fentanyl anesthesia. Anesthesiology. 1998 Jun;88(6):1459-66. doi: 10.1097/00000542-199806000-00007. PMID 9637637
- [Background] Nishina K, Mikawa K, Maekawa N, Obara H. Fentanyl attenuates cardiovascular responses to tracheal extubation. Acta Anaesthesiol Scand. 1995 Jan;39(1):85-9. doi: 10.1111/j.1399-6576.1995.tb05597.x. PMID 7725888
- [Background] Mendel P, Fredman B, White PF. Alfentanil suppresses coughing and agitation during emergence from isoflurane anesthesia. J Clin Anesth. 1995 Mar;7(2):114-8. doi: 10.1016/0952-8180(94)00024-x. PMID 7598918
- [Background] Sant'Ambrogio G, Widdicombe J. Reflexes from airway rapidly adapting receptors. Respir Physiol. 2001 Mar;125(1-2):33-45. doi: 10.1016/s0034-5687(00)00203-6. PMID 11240151
- [Background] Lema FE, Tafur LA, Giraldo C, Delgado MA. [Incidence of cough after desflurane and sevoflurane administration through a laryngeal mask: a controlled clinical trial]. Rev Esp Anestesiol Reanim. 2010 Mar;57(3):141-6. doi: 10.1016/s0034-9356(10)70188-2. Spanish. PMID 20422846
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Background] Grahame-Smith DG. How will knowledge of the human genome affect drug therapy? Br J Clin Pharmacol. 1999 Jan;47(1):7-10. doi: 10.1046/j.1365-2125.1999.00909.x. No abstract available. PMID 10073732
- [Background] Van Poucke GE, Bravo LJ, Shafer SL. Target controlled infusions: targeting the effect site while limiting peak plasma concentration. IEEE Trans Biomed Eng. 2004 Nov;51(11):1869-75. doi: 10.1109/TBME.2004.827935. PMID 15536889
- [Background] Tafur LA, Gómez JM, Parra LE. Validación de nomogramas de remifentanil y propofol para la administración de anestesia total endovenosa. Rev. Col. Anest. 2009; 37:21-8.
- [Background] Mertens MJ, Olofsen E, Engbers FH, Burm AG, Bovill JG, Vuyk J. Propofol reduces perioperative remifentanil requirements in a synergistic manner: response surface modeling of perioperative remifentanil-propofol interactions. Anesthesiology. 2003 Aug;99(2):347-59. doi: 10.1097/00000542-200308000-00016. PMID 12883407
- [Background] Eger EI 2nd. Age, minimum alveolar anesthetic concentration, and minimum alveolar anesthetic concentration-awake. Anesth Analg. 2001 Oct;93(4):947-53. doi: 10.1097/00000539-200110000-00029. PMID 11574362
- [Background] Matsuura T, Oda Y, Tanaka K, Mori T, Nishikawa K, Asada A. Advance of age decreases the minimum alveolar concentrations of isoflurane and sevoflurane for maintaining bispectral index below 50. Br J Anaesth. 2009 Mar;102(3):331-5. doi: 10.1093/bja/aen382. Epub 2009 Jan 24. PMID 19168857
- [Background] Albertin A, Casati A, Bergonzi P, Fano G, Torri G. Effects of two target-controlled concentrations (1 and 3 ng/ml) of remifentanil on MAC(BAR) of sevoflurane. Anesthesiology. 2004 Feb;100(2):255-9. doi: 10.1097/00000542-200402000-00012. PMID 14739797
- [Background] Olofsen E, Sleigh JW, Dahan A. The influence of remifentanil on the dynamic relationship between sevoflurane and surrogate anesthetic effect measures derived from the EEG. Anesthesiology. 2002 Mar;96(3):555-64. doi: 10.1097/00000542-200203000-00009. PMID 11873028
- [Background] Manyam SC, Gupta DK, Johnson KB, White JL, Pace NL, Westenskow DR, Egan TD. Opioid-volatile anesthetic synergy: a response surface model with remifentanil and sevoflurane as prototypes. Anesthesiology. 2006 Aug;105(2):267-78. doi: 10.1097/00000542-200608000-00009. PMID 16871060
- [Background] Dennis R. Cómo estimar el tamaño de la muestra en investigación con humanos. Acta Méd Colom. 1989;14: 92-99.
- [Background] Dobson AJ. Calculating simple size. Transactions of the Menzie Foundation. 1984; 7:75-79.
- [Background] Lerou JG. Nomogram to estimate age-related MAC. Br J Anaesth. 2004 Aug;93(2):288-91. doi: 10.1093/bja/aeh186. Epub 2004 Jun 25. PMID 15220181
- [Background] Coleridge HM, Coleridge JCC. Reflexes evoked from the tracheobronchial tree and lungs. In: Handbook of Physiology, Section 3: the Respiratory System, Vol II: Control of Breathing, Part I (Cherniack NS, Widdicombe JG, eds). Washington, DC:American Physiological Society, 1986;395-429.
- [Background] Widdicombe JG. Vagal reflexes in the airways. In: Neural Regulation of the Airways in Health and Disease (Kaliner M, Barnes PJ, eds). New York:Marcel Dekker, 1988;187-202.
- [Background] Lee DH, Park SJ. Effects of 10% lidocaine spray on arterial pressure increase due to suspension laryngoscopy and cough during extubation. Korean J Anesthesiol. 2011 Jun;60(6):422-7. doi: 10.4097/kjae.2011.60.6.422. Epub 2011 Jun 17. PMID 21738845
- [Background] Irwin RS. Complications of cough: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):54S-58S. doi: 10.1378/chest.129.1_suppl.54S. PMID 16428692
- [Background] Leech P, Barker J, Fitch W. Proceedings: Changes in intracranial pressure and systemic arterial pressure during the termination of anaesthesia. Br J Anaesth. 1974 Apr;46(4):315-6. doi: 10.1093/bja/46.4.315-a. No abstract available. PMID 4451611
- [Background] Lee B, Lee JR, Na S. Targeting smooth emergence: the effect site concentration of remifentanil for preventing cough during emergence during propofol-remifentanil anaesthesia for thyroid surgery. Br J Anaesth. 2009 Jun;102(6):775-8. doi: 10.1093/bja/aep090. Epub 2009 May 2. PMID 19411668
- [Background] Hohlrieder M, Tiefenthaler W, Klaus H, Gabl M, Kavakebi P, Keller C, Benzer A. Effect of total intravenous anaesthesia and balanced anaesthesia on the frequency of coughing during emergence from the anaesthesia. Br J Anaesth. 2007 Oct;99(4):587-91. doi: 10.1093/bja/aem203. Epub 2007 Jul 27. PMID 17660457
- [Background] Shajar MA, Thompson JP, Hall AP, Leslie NA, Fox AJ. Effect of a remifentanil bolus dose on the cardiovascular response to emergence from anaesthesia and tracheal extubation. Br J Anaesth. 1999 Oct;83(4):654-6. doi: 10.1093/bja/83.4.654. PMID 10673886
- [Background] Wilhelm W, Schlaich N, Harrer J, Kleinschmidt S, Muller M, Larsen R. Recovery and neurological examination after remifentanil-desflurane or fentanyl-desflurane anaesthesia for carotid artery surgery. Br J Anaesth. 2001 Jan;86(1):44-9. doi: 10.1093/bja/86.1.44. PMID 11575408
- [Background] Jun NH, Lee JW, Song JW, Koh JC, Park WS, Shim YH. Optimal effect-site concentration of remifentanil for preventing cough during emergence from sevoflurane-remifentanil anaesthesia. Anaesthesia. 2010 Sep;65(9):930-5. doi: 10.1111/j.1365-2044.2010.06450.x. PMID 20645945